CLINICAL TRIAL: NCT00508105
Title: Comparison of Two Methods of Fixation of Subscapularis During Shoulder Arthroplasty
Brief Title: Comparing Two Surgical Methods of Fixation of Subscapularis During Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHREB2006489-0H
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Subscapularis Peel; Morselized Osteotomy
Keywords: Osteoarthritis; Shoulder; subscapularis peel; osteotomy
MeSH Terms: conditions — Osteoarthritis | interventions — Osteotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- subscapularis peel (Active Comparator)
  Interventions: Procedure: subscapularis peel
- osteotomy (Active Comparator)
  Interventions: Procedure: osteotomy

INTERVENTIONS:
Procedure: subscapularis peel — Detachment of the subscapularis tendon from its insertion on the lesser tuberosity "the peel".
  Other Names: non applicable
  Arms: subscapularis peel
Procedure: osteotomy — This group will use a technique that involves elevation of the tendon with a wafer of bone in order to gain access to the shoulder.
  Other Names: non applicable
  Arms: osteotomy

SUMMARY:
This pilot study is being conducted to compare 2 methods of access to the shoulder for arthroplasty in patients with Osteoarthritis as we do not know has a better outcome.

DETAILED DESCRIPTION:
The study investigates the difference in disease specific quality of life between patients who undergo a subscapularis peel versus morselized osteotomy of the lesser tuberosity, as measured by the Western Ontario Osteoarthritis of the Shoulder (WOOS) at one year post-operatively in patients who undergo shoulder arthroplasty ?

ELIGIBILITY:
Inclusion Criteria:

* Patients who have failed standard non-surgical management of their shoulder arthritis who would benefit from a shoulder arthroplasty.

Exclusion Criteria:

* Active joint or systemic infection
* Significant muscle paralysis
* Rotator cuff tear arthroplasty
* Major medical illness
* Unable to speak or read English/French
* Psychiatric illness that precludes informed consent
* Unwilling to be followed for 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hosptial, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Lapner PL, Sabri E, Rakhra K, Bell K, Athwal GS. Healing rates and subscapularis fatty infiltration after lesser tuberosity osteotomy versus subscapularis peel for exposure during shoulder arthroplasty. J Shoulder Elbow Surg. 2013 Mar;22(3):396-402. doi: 10.1016/j.jse.2012.05.031. Epub 2012 Sep 1. PMID 22944077
- [Result] Lapner PL, Sabri E, Rakhra K, Bell K, Athwal GS. Comparison of lesser tuberosity osteotomy to subscapularis peel in shoulder arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2012 Dec 19;94(24):2239-46. doi: 10.2106/JBJS.K.01365. PMID 23318614

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subscapularis Peel | Osteotomy
Started | 44 | 43
Completed | 40 | 37
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subscapularis Peel | Osteotomy | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 11 | 38
  >=65 years | 17 | 32 | 49
Age, Continuous [Mean (Full Range); unit: years] | 70.4 [45 to 90] | 65.3 [34 to 85] | 67.8 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 18 | 16 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Subscapularis Strength
Description: Subscapularis muscle strength will be measured with an electronic handheld dynamometer. Patients are asked to press the dynamometer in towards their chest (belly-press) for a period of approximately 3 seconds before releasing. Strength is measured in kilograms of force.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Osteotomy | Subscapularis Peel
Number analyzed (Participants) | 43 | 44
kg | 4.4 (2.9) | 5.5 (2.6)

2. Secondary Outcome: Western Ontario Osteoarthritis of the Shoulder Index
Description: The Western Ontario Osteoarthritis of the Shoulder Index (WOOS) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WOOS is a patient-reported measure, 19-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.
Time Frame: 2 Years
Measure: Mean (Standard Deviation); unit: WOOS Score
Arm/Group | Osteotomy | Subscapularis Peel
Number analyzed (Participants) | 43 | 44
WOOS Score | 86.5 (16) | 88.2 (16.5)

3. Secondary Outcome: American Shoulder and Elbow Score
Description: The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Time Frame: 2 Years
Measure: Mean (Standard Deviation); unit: ASES Score
Arm/Group | Osteotomy | Subscapularis Peel
Number analyzed (Participants) | 43 | 44
ASES Score | 79.4 (24.6) | 83.3 (19)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through to participant study completion up until 2-years post-operative
Groups:
- Subscapularis Peel: tenotomy: This treatment group will undergo a technique that involves division of the tendon to gain access to the shoulder.
Arm/Group | Subscapularis Peel | Osteotomy
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No